CLINICAL TRIAL: NCT00988091
Title: A 26 Week, Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of Single Intra-Articular Injection 1.2% Sodium Hyaluronate for Treatment of Painful Osteoarthritis of the Knee, With Optional 26-Week Open-Label Safety Extension
Brief Title: Investigation of 1.2% Sodium Hyaluronate for Treatment of Painful Chronic Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-03
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Results first posted 2012-06-04 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IA-SA (Placebo Comparator): Each participant received a single intra-articular (IA) injection of buffered saline (SA) into the target knee, and was followed for a total of 26 weeks in the double-blind period. Participants had the option of continuing into the open-label period in which they could receive a single intra-articular injection of 1.2% sodium hyaluronate (IA-BioHA) into the target knee and be followed for an additional 26 weeks.
  Interventions: Device: Buffered Saline
- IA-BioHA (Experimental): Each participant received a single intra-articular (IA) injection of 1.2% sodium hyaluronate (BioHA) into the target knee, and was followed for a total of 26 weeks in the double-blind period. Participants had the option of continuing into the open-label period in which they received a single intra-articular injection of 1.2% sodium hyaluronate (IA-BioHA) into the target knee and were followed for an additional 26 weeks.
  Interventions: Device: 1.2% Sodium Hyaluronate

INTERVENTIONS:
Device: 1.2% Sodium Hyaluronate — IA-BioHA is supplied in a disposable 7 ml nominal volume glass syringe containing 60 mg/5 ml of 1.2% sodium hyaluronate. Participants are given a single injection in the target knee on Day 1 of the double-blind period and optionally on the first day of the open-label period (approximately week 27).
  Other Names: sodium hyaluronate
  Arms: IA-BioHA
Device: Buffered Saline — IA-SA is supplied in a disposable 7 ml nominal volume glass syringe containing 5 ml of phosphate buffered saline. Participants are given a single injection in the target knee on Day 1 of the double-blind period.
  Other Names: saline
  Arms: IA-SA

SUMMARY:
Subjects with chronic osteoarthritis of the knee will be assigned to receive an injection of either 1.2% sodium hyaluronate or buffered saline to evaluate its effectiveness and safety for 26 weeks. After 26 weeks, subjects can elect to receive a second injection of 1.2% sodium hyaluronate and be followed for another 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic osteoarthritis (OA) of target knee confirmed by American College of Rheumatology (ACR) Criteria.
* Pain due to OA in target knee present for at least 6 months.
* During Screening and Baseline visits, subjects will require a visual analog scale (VAS) score (100 mm) of ≥ 41 mm and ≤ 90 mm, recorded immediately following a 50-foot walk, AND at Baseline, cannot have decreased >10mm (improvement) from Screening.
* A bilateral standing anteroposterior (AP) X-ray confirming OA of the target knee.
* Ability and willingness to use only acetaminophen as the analgesic (rescue) study medication
* Ability to perform procedures required of the pain index evaluations (unassisted walking 50 feet on a flat surface and going up and down stairs).
* Willingness and ability to complete efficacy and safety questionnaires and ability to read and understand study instructions.
* Signed Subject Informed Consent Form

Exclusion Criteria:

* Any major injury (including sports injuries) to the target knee within the prior 12 months.
* Any surgery to the target knee, hip and contralateral hip within the prior 12 months.
* Major and minor articular procedures
* Inflammatory arthropathies such as rheumatoid arthritis, lupus arthropathy, or psoriatic arthritis.
* Gout or calcium pyrophosphate (pseudogout) diseases of the target knee that have flared within the previous 6 months.
* X-ray findings of acute fractures, severe loss of bone density, avascular necrosis, and/or severe bone or joint deformity in the target knee.
* Osteonecrosis of either knee.
* Fibromyalgia, pes anserine bursitis, lumbar radiculopathy, and/or neurogenic or vascular claudication.
* Significant anterior knee pain due to diagnosed isolated patella-femoral syndrome or chondromalacia in the target knee.
* Significant target knee joint infection or skin disorder/infection within the previous 6 months prior to study enrollment.
* Symptomatic OA of the hips, spine, or ankle, if it would interfere with the evaluation of the target knee.
* Known hypersensitivity to acetaminophen, sodium hyaluronate, or phosphate buffered saline solution.
* Women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period.
* Recurrent medical history of severe allergic or immune-mediated reactions or other immune disorders.
* Vascular insufficiency of lower limbs or peripheral neuropathy severe enough to interfere with the study evaluation.
* Current treatment or treatment within the previous 2 years prior to Screening for any malignancy unless specific written permission is provided by the Sponsor (excluding basal cell or squamous cell carcinoma of the skin).
* Chronic liver disease and active liver disease based on liver profile of aspartate aminotransferase (AST), alanine transaminase (ALT), and conjugated bilirubin >2 times the upper limit of normal.
* Renal insufficiency based on serum creatinine >2.0 mg/dL.
* Any clinically significant laboratory value based on clinical history that the Investigator feels may affect the study evaluation.
* Any intercurrent chronic disease or condition that may interfere with the completion of the 6-month (or 12-month) follow-up of the study, such as liver disease, severe coronary disease, drug abuse, disordered mental state, or other clinically significant condition.
* Current alcoholism, and/or any known current addiction to pain medications.
* Any clinically significant finding that would place the patient at health risk, impact the study, or affect the completion of the study.
* Any psychiatric illness that would prevent comprehension of the details and nature of the study.
* Participation in any experimental device study within 6 months prior to the Screening, or an experimental drug study within 1 month prior to the Screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (34):
- United States (34):
  - Apex Clinical Trials, LLC, Homewood, Alabama
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - St. Joseph's Mercy Clinic, Hot Springs, Arkansas
  - Rx Medical Research of Arkansas, Inc, Little Rock, Arkansas
  - Southbay Pharma Research, Buena Park, California
  - Providence Clinical Research, Burbank, California
  - Triwest Research Associates, La Mesa, California
  - UCLA-Division of Rheumatology, Los Angeles, California
  - Investigational Site, Santa Barbara, California
  - Colorado Arthritis Center, PC, Englewood, Colorado
  - Front Range Clinical Research, Wheat Ridge, Colorado
  - New England Research Associates, LLC, Trumball, Connecticut
  - International Physicians Research, Aventura, Florida
  - Investigational Site, Fort Lauderdale, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - Tri-County Orthopaedic Center, Leesburg, Florida
  - Clinical Research Center LLC, Wellington, Florida
  - National Pain Research Institute, LLC, Winter Park, Florida
  - Georgia Institute for Clinical Research, Marietta, Georgia
  - Pinnacle Orthopaedics and Sports Medicine, Marietta, Georgia
  - Lee Research Institute, Shawnee, Kansas
  - Professional Research Network of Kansas, Wichita, Kansas
  - New Jersey Physicians, LLC, Passaic, New Jersey
  - Research Department, Bone & Joint Hospital at St. Anthony, Oklahoma City, Oklahoma
  - Omega Medical Research, Warwick, Rhode Island
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Palmetto Clinical Trial Services, LLC, Simpsonville, South Carolina
  - Black Hills Orthopedic & Spine Center, Rapid City, South Dakota
  - Holston Medical Group, Kingsport, Tennessee
  - McKenzie Medical Center, McKenzie, Tennessee
  - Texas Orthopedic Specialists, PA, Grapevine, Texas
  - Memorial Bone & Joint Research Foundation, Houston, Texas
  - Discovery Clinical Trials (DCT) - Stone Oak, LLC, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1007 subjects were screened for the double-blind period of the study, and 596 subjects were randomized and treated (safety population).
Period: Double-blind Period
Arm/Group | IA-SA | IA-BioHA
Started | 298 | 298
Intent to Treat Population | 294 (ITT population excludes participants from one site which was closed for non-compliance.) | 295 (ITT population excludes participants from one site which was closed for non-compliance.)
Completed | 255 | 251
Not Completed | 43 | 47
Not completed — Withdrawal by Subject | 15 | 13
Not completed — Lost to Follow-up | 12 | 14
Not completed — Other | 8 | 8
Not completed — Adverse Event | 6 | 9
Not completed — Use of exclusionary medication | 2 | 3
Period: Open-label Period
Arm/Group | IA-SA | IA-BioHA
Started | 229 (Participation in the Open-label period was optional.) | 225 (Participation in the Open-label period was optional.)
Completed | 208 | 192
Not Completed | 21 | 33
Not completed — Adverse Event | 4 | 7
Not completed — Use of exclusionary medication | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 10 | 16
Not completed — Lost to Follow-up | 3 | 5
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IA-SA | IA-BioHA | Total
Number analyzed (Participants) | 298 | 298 | 596
Age Continuous [Mean (Standard Deviation); unit: years] | 60.30 (11.180) | 60.70 (10.228) | 60.50 (10.708)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193 | 168 | 361
  Male | 105 | 130 | 235

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Visual Analogue Score (VAS) Pain Score of the 50-foot Walk Test at Week 26
Description: The level of pain is estimated by the participant following a walk of 50 feet in length which is observed by the investigator. Pain estimates were recorded on a 100 millimeter visual analog scale. A score of 0 millimeters means there was no pain; a score of 100 millimeters means extreme pain. Change from baseline is calculated: week 26 VAS Pain Score - Baseline VAS Pain Score.
Time Frame: Day 0 (baseline) through Week 26
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IA-SA | IA-BioHA
Number analyzed (Participants) | 294 | 295
units on a scale | -33.48 (1.81) | -28.15 (1.82)
Statistical Analysis 1: Comparison: IA-SA vs IA-BioHA; A treatment difference of >=7.0 mm and a pooled SD of 27.6 mm, requires a sample size of 244 subjects/treatment to complete the trial at 80% power at a two-sided significance level of 5%. To account for 18% dropout rate, the sample size was increased to 298/arm (total of 596). The primary null hypothesis (Ho) is that the effect of the two treatment groups at 26 weeks is equal and the corresponding alternative hypothesis (HA) is that the effect of the two treatment groups at 26 weeks is unequal; Test type: Superiority or Other; p = 0.034, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons because there was a single treatment comparison for the primary endpoint. The a priori threshold for statistical significance was p <0.05; The analysis included baseline score as a covariate and study center as a stratification variable; Adjusted mean difference = 5.33, 95% CI 2-sided [0.41 to 10.24]

2. Secondary Outcome: Change From Baseline in Western Ontario McMaster University Osteoarthritis Index (WOMAC) Disability Scores at Week 26
Description: Adjusted mean of all WOMAC pain, stiffness and physical function subscores on Visual Analog Scale (VAS) of 100 mm; 0 mm = no pain, stiffness and difficulty; 100 mm = extreme pain, stiffness and difficulty. Change from baseline calculated as: Week 26 minus baseline.
Time Frame: Day 0 (baseline), week 26
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IA-SA | IA-BioHA
Number analyzed (Participants) | 294 | 295
units on a scale | -21.72 (1.55) | -18.82 (1.57)
Statistical Analysis 1: Comparison: IA-SA vs IA-BioHA; The null hypothesis (Ho) is that the effect of the two treatment groups at 26 weeks is equal and the corresponding alternative hypothesis (HA) is that the effect of the two treatment groups at 26 weeks is unequal; Test type: Superiority or Other; p = 0.175, Mixed Models Repeated Measures ANCOVA — For secondary outcome measures, fixed-sequence testing was used in a sequentially rejective fashion. The a priori threshold for statistical significance was p <0.05; The analysis included baseline score as a covariate and study center as a stratification variable; Adjusted mean difference = 2.89, 95% CI 2-sided [-1.29 to 7.08]

3. Secondary Outcome: Percentage of Participants With a >=20mm Improvement Between Baseline and Week 26 on the 50 Foot Walk Visual Analogue Scale (VAS) Pain Score.
Description: The level of pain is estimated by the participant following a walk of 50 feet in length which is observed by the investigator. Pain estimates were recorded on a 100 millimeter visual analog scale. A score of 0 millimeters means there was no pain; a score of 100 millimeters means extreme pain. Change from baseline is calculated: week 26 VAS Pain Score - Baseline VAS Pain Score. The percent of participants who showed a 20mm or greater improvement in the pain scores at week 26 compared to baseline are reported.
Time Frame: Day 0 (baseline), Week 26
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | IA-SA | IA-BioHA
Number analyzed (Participants) | 256 | 253
percentage of participants | 66.8 | 60.9
Statistical Analysis 1: Comparison: IA-SA vs IA-BioHA; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.193, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; The analysis included study center as a stratification variable; Odds Ratio (OR) = 0.777, 95% CI 2-sided [0.532 to 1.136]

4. Secondary Outcome: Subjective Patient Assessment of Treatment at Week 26
Description: At the end of the double-blind period (week 26), participants were asked: "Are you satisfied with the results of the injection?" Answers could be: 1=dissatisfied; 2=slightly satisfied; 3=satisfied; or 4=very satisfied.
Time Frame: Week 26
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IA-SA | IA-BioHA
Number analyzed (Participants) | 266 | 269
units on a scale | 2.71 (1.096) | 2.70 (1.115)
Statistical Analysis 1: Comparison: IA-SA vs IA-BioHA; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.887, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; The analysis included study center as a stratification variable

5. Secondary Outcome: Number of Tablets of Rescue Medication Used Between Visits
Description: Acetaminophen (500-mg tablets) was provided to study participants as a rescue medication in case they needed a pain medication during the study. The mean number of tablets of rescue medication should have been summarized, however the data was not captured in a reliable way and is therefore not reported.
Time Frame: Day 1 to week 26
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | IA-SA | IA-BioHA
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Patient Global Assessment at Week 26
Description: Participants were asked to mark along a 100mm visual analog scale (VAS) indicating the point best representing the severity of the knee pain that day. The left side of the VAS was 0=no pain and the right side was 100 = extreme pain. Change from baseline was calculated as Week 26 - Baseline.
Time Frame: Day 0 (baseline), Week 26
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IA-SA | IA-BioHA
Number analyzed (Participants) | 294 | 295
units on a scale | -27.41 (1.83) | -23.41 (1.85)
Statistical Analysis 1: Comparison: IA-SA vs IA-BioHA; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.116, Mixed Models Repeated Measures ANCOVA — [p-value comment as in outcome 2, analysis 1]; The analysis included baseline score as a covariate and study center as a stratification variable; Adjusted mean difference = 4.00, 95% CI 2-sided [-0.99 to 8.98]

7. Secondary Outcome: Percentage of Observed Osteoarthritis Research Society International (OARSI30) Responders Using the Visual Analogue Scale (VAS) to Assess Pain Following a 50-foot Walk at Week 26
Description: Responders are identified based on a calculation of three scales: 50-foot walk test for pain, function (WOMAC Disability score) and global assessment (Patient Global Assessment Score) scales. Each of the individual scales was completed by the participant. A responder showed considerable improvement in pain or function (>=50 percent and absolute change of >=20 millimeters), or improvement in at least two of three categories: Pain and/or Function and/or Patient Global Assessment scales of >=20 percent and absolute change >=10 millimeter. Response at Week 26 is compared to baseline.
Time Frame: Day 0 (baseline), week 26
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | IA-SA | IA-BioHA
Number analyzed (Participants) | 253 | 249
percentage of participants | 70.0 | 62.2
Statistical Analysis 1: Comparison: IA-SA vs IA-BioHA; The null hypothesis (Ho) is that the effect of the two treatment groups at 26 weeks is equal and the corresponding alternative hypothesis (HA) is that the effect of the two treatment groups at 26 weeks is unequal.[; Test type: Superiority or Other; p = 0.081, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; The analysis included study center as a stratification variable; Odds Ratio (OR) = 0.710, 95% CI 2-sided [0.483 to 1.044]

ADVERSE EVENTS:
Time Frame: Double-blind period is day 1 to week 26. The open-label period is week 27 to week 52.
Groups:
- IA-SA: Double-blind Period: Each participant received a single intra-articular (IA) injection of buffered saline (SA) into the target knee, and was followed for a total of 26 weeks in the double-blind period.
- IA-BioHA: Double-blind Period: Each participant received a single intra-articular (IA) injection of 1.2% sodium hyaluronate (BioHA) into the target knee, and was followed for a total of 26 weeks in the double-blind period.
- IA-BioHA: Open-label Period: Participants had the option of continuing into the open-label period in which their target knee received a single intra-articular (IA) injection of 1.2% sodium hyaluronate (BioHA) and they were followed for an additional 26 weeks.
Arm/Group | IA-SA: Double-blind Period | IA-BioHA: Double-blind Period | IA-BioHA: Open-label Period
Serious Adverse Events (participants affected / at risk) | 6/298 | 13/298 | 12/454
Other Adverse Events (participants affected / at risk) | 25/298 | 29/298 | 32/454
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IA-SA: Double-blind Period (N=298) | IA-BioHA: Double-blind Period (N=298) | IA-BioHA: Open-label Period (N=454)
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Myopericarditis (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Urethral intrinsic sphincter deficiency (Congenital, familial and genetic disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0
Intraspinal abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Heart rate irregular (Investigations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Nephrectomy (Surgical and medical procedures) | 0 | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IA-SA: Double-blind Period (N=298) | IA-BioHA: Double-blind Period (N=298) | IA-BioHA: Open-label Period (N=454)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 29 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.